CLINICAL TRIAL: NCT05517135
Title: tReatment Individualisation By EBV stratificatiON in Nasopharyngeal Carcinoma: an Umbrella Platform Study (RIBBON-Umbrella)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/2315
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; EBV DNA; Biomarker-guided; Treatment Individualization; Risk Stratification
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — DMAC2L protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tissue, fresh tumour biopsy tissue, saliva and peripheral blood samples will be obtained for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Arm 1: Arm 1: Pre-treatment EBV DNA <4000 copies/mL AND N0-1 or T4N0 (TNM AJCC/UICC 8th edition)
  Interventions: Other: Arm 1
- Arm 2: Arm 2: Pre-treatment EBV DNA ≥4000 copies/mL OR N2-N3 OR T4N+ (TNM AJCC/UICC 8th edition) AND EBV DNA UNDETECTABLE after 2-3 cycles of induction chemotherapy (IC)
  Interventions: Other: Arm 2
- Arm 3: Arm 3: Pre-treatment EBV DNA ≥4000 copies/mL OR N2-N3 OR T4N+ (TNM AJCC/UICC 8th edition) AND EBV DNA DETECTABLE after 2-3 cycles of IC
  Interventions: Other: Arm 3
- Group 1: Group 1: Recurrent/metastatic NPC, EBV DNA <4000 copies/mL
  Interventions: Other: Group 1
- Group 2: Group 2: Recurrent/metastatic NPC, EBV DNA ≥4000 copies/mL
  Interventions: Other: Group 2

INTERVENTIONS:
Other: Arm 1 — Concurrent chemoradiotherapy (CCRT) using cisplatin (100 mg/m2 IV) or carboplatin (AUC 5 IV) with radiotherapy +/- adjuvant chemotherapy (AC). For AC, physicians can choose between cisplatin-5FU d1-4, q4w for 3 cycles, or capecitabine 650 mg/m2 bid for 12 months or 1000 mg/m2 bid oral, d1-21, q3w for 6 months
  Groups: Arm 1
Other: Arm 2 — IC using cisplatin (80 mg/m2 IV) or carboplatin (AUC 3-5 IV) in combination with gemcitabine (1000 mg/m2 d1,8) or 5-fluorouracil (1000 mg/m2 bolus IV d1-4) or docetaxel (75 mg/m2 IV), and CCRT +/- metronomic capecitabine (650 mg/m2 bid oral for 12 months)
  Groups: Arm 2
Other: Arm 3 — IC using cisplatin (80 mg/m2 IV) or carboplatin (AUC 3-5 IV) in combination with gemcitabine (1000 mg/m2 d1,8) or 5-fluorouracil (1000 mg/m2 bolus IV d1-4) or docetaxel (75 mg/m2 IV), followed by either of the following:
  1. RIBBON-LA-01 (NCT06093061)
  2. CCRT + metronomic capecitabine (650 mg/m2 bid oral for 12 months)
  Groups: Arm 3
Other: Group 1 — Combination chemotherapy (using cisplatin or carboplatin with gemcitabine, 5-fluorouracil or docetaxel) and consolidative RT to the nasopharynx and neck (if good response to chemotherapy) +/- metastasis-directed therapy (surgery, radiofrequency ablation or RT) +/- immune checkpoint blockade (ICB) or capecitabine
  Groups: Group 1
Other: Group 2 — Combination chemotherapy (using cisplatin or carboplatin with gemcitabine, 5-fluorouracil or docetaxel) with or without ICB +/- maintenance ICB or capecitabine
  Groups: Group 2

SUMMARY:
This is a prospective platform study that will investigate the outcomes of patients with locoregionally-advanced nasopharyngeal carcinoma (LA-NPC) or recurrent-metastatic nasopharyngeal carcinoma (RM-NPC) who are assigned to treatment arms of different chemotherapy sequencing and intensity based on their pre- and on-treatment plasma EBV DNA results.

DETAILED DESCRIPTION:
The primary objectives of this platform are: (1) to prospectively validate the prognostic potential of an EBV DNA-based risk-stratification strategy of patients with LA- and RM-NPC; and (2) to test if treatment individualization strategies based on pre- and on-treatment plasma EBV DNA will improve survival outcomes.

For LA-NPC, the study design consists of two components: (1) to allocate adult patients with UICC/AJCC 8th edition TNM-stage 2-4A LA-NPC to 3 treatment arms of different intensities by their plasma EBV DNA levels pre-treatment and post-induction chemotherapy (IC); and (2) to incorporate open-label, single-arm, phase 2 trials within the platform for patients who are deemed to be at high-risk of relapse, defined by a persistently detectable EBV DNA following 3 cycles of IC. Primary study end-point is 2-year disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

Each patient eligible to participate in this study must meet all the following criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Age ≥21 years on the day of signing the ICF
3. Fulfil one of the following three scenarios:

   1. Suspected NPC cases, diagnosed clinically based on symptoms (neck swelling, unilateral epistaxis, nasal obstruction etc.)
   2. Newly-diagnosed, histologically confirmed NPC patients with Stages 2-4A disease based on the AJCC/UICC 8th Edition TNM stage classification
   3. Newly-diagnosed patients with RM-NPC

   All confirmed NPC patients must meet these additional criteria before they can continue participation in the study:
4. NPC associated with EBV infection, determined as:

   1. The presence of EBV has been confirmed in the tumour by immunohistochemistry for EBV antigens or in situ hybridization for EBV early RNA (EBER), or
   2. NPC occurred in association with a raised serum titre of IgA to EBV viral capsid antigen (VCA) or early antigen (EA) in a patient living in endemic area of high incidence of EBV+ undifferentiated NPC, or
   3. NPC in the context of an elevated circulating EBV genome level
5. AJCC 8th edition stage 2-4A or RM NPC based on the following diagnostic workup:

   1. Evaluation of tumour extent with magnetic resonance imaging (MRI) of the nasopharynx and neck. If MRI is medically contraindicated, computed tomography (CT) scan with ≤3 mm and intravenous contrast is acceptable.
   2. Distant metastasis staging:

      * CT scan with contrast of the chest, abdomen, and pelvis or a total body 18F-Fluorodeoxygenase positron emission tomography CT (18F-FDG-PET-CT) scan;
      * Bone scan, if a 18F-FDG-PET-CT scan is not performed.
6. ECOG Performance Status ≤1
7. Adequate organ function

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to enrol:

1. Age <21 years or >99 years old
2. Has received any prior RT or systemic anti-cancer therapy including investigational agents that are not part of the intended treatment plan for NPC
3. Any known central nervous system metastases and/or carcinomatous meningitis
4. Any active malignancy ≤2 years before start of study except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
5. Patients with severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.

   a. Severe infections within 4 weeks before start of study, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
6. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is >500 IU/mL or patients with active hepatitis C virus (HCV) should be excluded.

   Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA <500 IU/mL), and cured hepatitis C patients can be enrolled
7. Prior allogeneic stem cell transplantation or organ transplantation
8. Any of the following cardiovascular risk factors:

   1. Cardiac chest pain, defined as moderate pain or any cardiac condition e.g., arrhythmias, malignant hypertension, etc. that limits instrumental activities of daily living, ≤28 days before start of study
   2. Pulmonary embolism ≤28 days before start of study
   3. Any history of cerebrovascular accident or seizure ≤ 28 days before start of study
9. A history of severe hypersensitivity reactions to gemcitabine, cisplatin, capecitabine and/or any of its excipients
10. Has received any herbal medicine used to control cancer within 14 days of the start of study
11. Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for adverse events (AEs) not considered a likely safety risk (eg, alopecia, neuropathy and specific laboratory abnormalities)
12. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of treatment or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct
13. Concurrent participation in another therapeutic clinical study

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected NPC or histologically confirmed NPC will be recruited for the study. Patients with confirmed stage 2-4B NPC will be enrolled into the platform study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 2 years from end of treatment

SECONDARY OUTCOMES:
Overall survival | 2 years after end of treatment
Distant metastasis-free survival | 2 years after end of treatment
Loco-regional recurrence-free survival | 2 years after end of treatment
Treatment-related adverse events | From start of treatment to 30 days after last treatment and up to 5 years post - treatment
Genome sequencing of biological samples | baseline, mid/post IC, mid CCRT, 1-2 weeks post-RT, 3 months post-RT/mid-adjuvant chemotherapy, at point of recurrence and post immune checkpoint blockade treatment (for recurrence, if any) up to 5 years
  Blood samples will be collected at up to 7 timepoints - baseline, mid/post IC, mid CCRT, 1-2 weeks post-RT, 3 months post-RT/mid-adjuvant chemotherapy, at point of recurrence and post immune checkpoint blockade treatment (ICB) for recurrence, if any; fresh biopsy samples will be collected at baseline, mid-IC, at point of recurrence and mid-ICB, if amenable for biopsy. Saliva samples will be collected at baseline and at point of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Lee Kiang Chua, MBBS, FRCR, PhD, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore